CLINICAL TRIAL: NCT04746794
Title: Implementing the Moon: Getting Genomic Testing to the Public
Brief Title: Early Detection of GEnetic Risk (EDGE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elizabeth Swisher, Gynecologic oncologist, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00009476; 1U01CA232795-01A1 (NIH); RG1123410 (Registry Identifier: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-12-29; First posted 2021-02-10 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Genetic Predisposition
Keywords: Primary Care; Genetic Testing; Risk Assessment; Hereditary Cancer; Implementation
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Point of Care (Experimental): For clinics in the point of care (POC) arm, patients will be approached at the time they come in to the clinic for a routine visit with their primary care provider. We will screen patients for familial cancer risk using electronic tablets in the waiting room or, in the case of a telehealth visit, through telephone contact before the visit. Patients identified as high risk will be offered genetic testing for a panel of hereditary cancers.
  Interventions: Behavioral: Population-level screening
- Direct Patient Engagement (Experimental): For clinics in the direct patient engagement (DPE) arm, patients will be identified by reviewing clinic records to create an "active" patient list (i.e., those who have had a visit in the past year). We will contact patients by postal mail and email to provide a link to the online risk screening tool. The patient outreach is not tied to a specific visit and the online screening can be completed at any time. Patients identified as high risk will be offered genetic testing for a panel of hereditary cancers.
  Interventions: Behavioral: Population-level screening
- Stakeholder Interviews and Surveys (No Intervention): Samples of patients, providers, and clinic leaders will be assessed at several points throughout the study - baseline and follow-up. We will use a mixed methods approach, with both quantitative assessments (surveys) and qualitative assessments (interviews). Baseline assessments will provide initial data on the patient population and current clinic functioning and help in implementation planning. The final assessments will provide estimates of change in patients, providers, and clinic leaders as a result of the implementation.

INTERVENTIONS:
Behavioral: Population-level screening — The study intervention involves having patients complete a familial cancer risk assessment survey. Those who are found to be at high risk will be offered genetic testing for a panel of hereditary cancers. A "previvor" plan will be created to assist patients and their providers in completing the appropriate follow-up for those with a mutation identified.
  Arms: Direct Patient Engagement; Point of Care

SUMMARY:
The study intervention involves having patients complete a familial cancer risk assessment survey. Those who are found to be at high risk will be offered genetic testing for a panel of hereditary cancers. A "previvor" plan will be created to assist patients and their providers in completing the appropriate follow-up for those with a mutation identified.

DETAILED DESCRIPTION:
Current practice guidelines from ACMG (American College of Medical Genetics and Genomics) provide referral indications for cancer predisposition assessment. Identifying patients with high genetic risk for breast, ovary, colon, or other cancers has important clinical ramifications for an individual's healthcare, but genetic risk if often not identified because of testing barriers at several levels. Barriers at the provider level include inadequacies in risk recognition, patient referrals and availability of genetic professionals to provide counseling in a traditional testing paradigm. Barriers at the level of the patient include poor understanding of the availability and benefits of testing and inadequate access to testing services. How to best implement appropriate genomic testing and follow-up care into an operating healthcare system is not known. Issues of communication, clinical flow, reportable actions, and transmission of information and support are of critical importance, and must change and grow to accommodate the new information contained within genomic testing. Studies to date of the implementation process have been conducted in high resourced facilities, under optimal conditions, often not at the system level. Aims include:

1. Compare the efficacy and implementation of two strategies for identifying members of a primary care clinic's population who have a family or personal history of cancer and offering high-risk individuals to obtain genetic testing for cancer susceptibility mutations in a randomized trial. The two methods are: 1) Point of Care (POC) approach: A tablet-based screening for family/personal history of cancer will be offered to all patients aged 25 and up coming in for a routine appointment at the clinic. 2) Direct Patient Engagement (DPE): Emails and letters will be sent to all individuals aged 25 and older in a clinic's population, inviting them to visit a web site for screening for family /personal history of cancer. In both strategies, those determined to be high-risk will receive online education about genetic testing and an invitation to obtain such testing through a web-based platform. Randomization will occur at the clinic level, with half of the clinics using the POC approach and the other half using DPE. Outcomes will be the fraction of the active clinic patient population that completes screening and the fraction of the active clinic patient population that undergoes testing.

   Hypothesis 1: DPE screening will result in a higher proportion of active patients who screen for familial cancer risk compared with POC screening.

   Hypothesis 2: Of screened patients, POC patients will produce a higher proportion of tested patients compared with DPE.
2. Identify changes, problems, and inefficiencies in clinical flow and interactions during and after the implementation of genomic testing for cancer risk across primary care clinics.
3. Evaluate the effects of two methods of implementation of genomic screening for cancer risk on patient, provider, and health system leader reports of benefits and harms, satisfaction, perceived quality of care, including across gender, racial/ethnic, socioeconomic, and genetic literacy divides.
4. Evaluate the value (cost-effectiveness) and affordability (budget impact) of each screening strategy.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Age 25 or older
* An active patient at a participating clinic (had at least one visit in the past 12 months)
* Comfortable reading and writing in English

Exclusion Criteria:

* Those who do not meet inclusion criteria.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20184 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Swisher, MD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Billings Clinic, Billings, Montana
  - MultiCare Health System, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swisher EM, Harris HM, Knerr S, Theoryn TN, Norquist BM, Brant J, Shirts BH, Beers F, Cameron D, Dusic EJ, Riemann LA, Devine B, Raff ML, Kadel R, Cabral HJ, Wang C. Strategies to Assess Risk for Hereditary Cancer in Primary Care Clinics: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2025 Mar 3;8(3):e250185. doi: 10.1001/jamanetworkopen.2025.0185. PMID 40053353

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 primary care clinics (units) were randomized to use one of two engagement strategies. Patients who had an appointment at a clinic randomized to the POC arm were approached using the POC strategy (described below). Patients seen at a DPE clinic were approached using the DPE strategy. Recruitment began in September of 2020 and ended in February of 2023.
Pre-assignment Details: As randomization was done by clinic, 115,484 individuals started the study (115,319 patients; 165 primary care providers). The 95,623 patients seen during the 12 month window set by the study protocol serve as the denominator for the main outcomes (proportion of patients who completed the cancer risk assessment screening; proportion of patients who completed genetic testing). 20,184 individuals were officially enrolled through completing surveys or the cancer risk assessment screening.
Units Other Than Participants: Clinics
Groups:
- Point of Care: Clinics in the point of care (POC) arm approached patients at the time they came in to the clinic for a routine visit with their primary care provider. The familial cancer risk screening was completed using electronic tablets in the waiting room or, in the case of a telehealth visit, through telephone contact before the visit. Patients identified as likely to benefit based on their risk profile, were offered genetic testing for a panel of hereditary cancers.
- Direct Patient Engagement: Clinics in the direct patient engagement (DPE) arm contacted patients by postal mail and email to provide a link to the online familial cancer risk screening tool. This occurred one to three months after the patient had a routine visit with their primary care provider. Patients identified as likely to benefit based on their risk profile, were offered genetic testing for a panel of hereditary cancers.
Period: Overall Study
Arm/Group | Point of Care | Direct Patient Engagement
Started | 63820; 6 Clinics | 51664; 6 Clinics
Patients With a Primary Care Visit | 63750; 6 Clinics | 51664; 6 Clinics
Clinic Primary Care Providers and Clinic Leaders | 70; 6 Clinics | 95; 6 Clinics
Completed Surveys Only (Providers and Clinic Leaders) (not part of outcome measures) | 46; 6 Clinics | 37; 6 Clinics
Completed Surveys Only (Patients) (not part of outcome measures) | 2323; 6 Clinics | 2272; 6 Clinics
Completed Cancer Risk Screening (Patients) | 11148; 6 Clinics | 4358; 6 Clinics
TOTAL ENROLLED | 13517; 6 Clinics | 6667; 6 Clinics
Patients With a Primary Care Visit During 12m Study Window (Denominator for Outcome Measures) | 51693; 6 Clinics | 43930; 6 Clinics
Health System A - Patients in 12m Study Window (Only data from Health System A is used in Outcomes 3-5) | 29862; 3 Clinics | 21457; 3 Clinics
Completed Cancer Risk Screening During 12m Study Window | 9892; 6 Clinics | 3813; 6 Clinics
Eligible for Genetic Testing | 3070; 6 Clinics | 1603; 6 Clinics
Completed Genetic Testing | 757; 6 Clinics | 717; 6 Clinics
Completed | 13517; 6 Clinics | 6667; 6 Clinics
Not Completed | 50303; 0 Clinics | 44997; 0 Clinics
Not completed — Did not complete any study assessment | 50303 | 44997

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are provided for all patients who completed the cancer risk assessment screening. And for patients and primary care providers who completed a baseline survey prior to study launch. Patients, Providers, and Clinic Leaders who enrolled in the study by completing surveys post-intervention did not have Baseline data collected (2,286).
Units Other Than Participants: Clinics
Groups:
- Total: Total of all reporting groups
Arm/Group | Point of Care | Direct Patient Engagement | Total
Number analyzed (Participants) | 12316 | 5582 | 17898
Number analyzed (Clinics) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Primary Care Providers and Clinic Leaders were not asked for their age.
  years
    Patients who completed cancer risk assessment screening: number analyzed (Participants) | 11148 | 4358 | 15506
    Patients who completed cancer risk assessment screening | 59.0 (16.2) | 58.0 (14.9) | 58.9 (15.1)
    Patients who completed a baseline survey: number analyzed (Participants) | 1128 | 1191 | 2319
    Patients who completed a baseline survey | 61.7 (15.2) | 61.0 (15.3) | 61.3 (15.3)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Analysis for Patients is listed separately from Providers and Clinic Leaders.
  Participants
    Female (Patients): number analyzed (Participants) | 12276 | 5549 | 17825
    Female (Patients) | 7359 | 3834 | 11193
    Male (Patients): number analyzed (Participants) | 12276 | 5549 | 17825
    Male (Patients) | 4481 | 1693 | 6174
    Unknown (Patients): number analyzed (Participants) | 12276 | 5549 | 17825
    Unknown (Patients) | 436 | 22 | 458
    Female (Providers and Clinic Leaders): number analyzed (Participants) | 40 | 33 | 73
    Female (Providers and Clinic Leaders) | 21 | 16 | 37
    Male (Providers and Clinic Leaders): number analyzed (Participants) | 40 | 33 | 73
    Male (Providers and Clinic Leaders) | 12 | 10 | 22
    Unknown (Providers and Clinic Leaders): number analyzed (Participants) | 40 | 33 | 73
    Unknown (Providers and Clinic Leaders) | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity was NOT asked of patients who completed the cancer risk assessment screening.
  Participants
    Patients: number analyzed (Participants) | 1128 | 1191 | 2319
    Patients: Hispanic or Latino | 21 | 37 | 58
    Patients: Not Hispanic or Latino | 997 | 1046 | 2043
    Patients: Unknown or Not Reported | 110 | 108 | 218
    Providers and Clinic Leaders: number analyzed (Participants) | 40 | 33 | 73
    Providers and Clinic Leaders: Hispanic or Latino | 1 | 2 | 3
    Providers and Clinic Leaders: Not Hispanic or Latino | 30 | 23 | 53
    Providers and Clinic Leaders: Unknown or Not Reported | 9 | 8 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race was NOT asked of patients who completed the cancer risk assessment screening.
  Participants
    Patients: number analyzed (Participants) | 1128 | 1191 | 2319
    Patients: American Indian or Alaska Native | 7 | 11 | 18
    Patients: Asian | 21 | 31 | 52
    Patients: Native Hawaiian or Other Pacific Islander | 4 | 2 | 6
    Patients: Black or African American | 14 | 17 | 31
    Patients: White | 1000 | 1037 | 2037
    Patients: More than one race | 33 | 38 | 71
    Patients: Unknown or Not Reported | 49 | 55 | 104
    Providers and Clinic Leaders: number analyzed (Participants) | 40 | 33 | 73
    Providers and Clinic Leaders: American Indian or Alaska Native | 0 | 0 | 0
    Providers and Clinic Leaders: Asian | 2 | 4 | 6
    Providers and Clinic Leaders: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Providers and Clinic Leaders: Black or African American | 0 | 0 | 0
    Providers and Clinic Leaders: White | 31 | 20 | 51
    Providers and Clinic Leaders: More than one race | 0 | 3 | 3
    Providers and Clinic Leaders: Unknown or Not Reported | 7 | 6 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12316 | 5582 | 17898

OUTCOME MEASURES:

1. Primary Outcome: Rates of Screening
Description: Fraction of the active clinic patient population that completed screening
Time Frame: 1 year
Population: Patients 25 years of age or older, comfortable speaking English, who had an appointment at one of the participating clinics during the 12 month recruitment window.
Measure: Count of Participants; unit: Participants
Arm/Group | Point of Care | Direct Patient Engagement
Number analyzed (Participants) | 51693 | 43930
Participants | 9892 | 3813
Statistical Analysis 1: Comparison: Point of Care vs Direct Patient Engagement; Test type: Superiority; p = 0.0074, Chi-squared

2. Primary Outcome: Rates of Testing
Description: Fraction of the active clinic patient population that completed genetic testing.
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Point of Care | Direct Patient Engagement
Number analyzed (Participants) | 51693 | 43930
Participants | 757 | 717
Statistical Analysis 1: Comparison: Point of Care vs Direct Patient Engagement; Test type: Superiority; p < 0.0001, Chi-squared

3. Secondary Outcome: Total Cost of Each Engagement Strategy
Description: This outcome is the total costs for each engagement strategy, scaled to a healthcare system of 100,000 patients. The total costs from the health-system perspective is the sum of program costs and staff costs over 2 years, in U.S. dollars. The cost from the limited societal perspective includes patient costs in addition to health-system costs. The total costs will be used in the incremental cost calculation below.
Time Frame: 2 years
Population: Data from only one of the participating healthcare systems were used. There were 3 clinics in the POC arm and 3 clinics in the DPE arm. Costs were calculated at the per-patient level and scaled to apply to a theoretical healthcare system with 100,000 patients.
Measure: Number; unit: cost in $
Arm/Group | Point of Care | Direct Patient Engagement
Number analyzed (Participants) | 29,862 | 21,457
cost in $
  Cost from health-system perspective | 640,776 | 697,116
  Cost from limited societal perspective (includes patient costs) | 648,395 | 698,350

4. Secondary Outcome: Incremental Cost When Comparing Two Engagement Strategies
Description: This outcome is the comparative (incremental) cost of two different engagement strategies for population-based risk assessment for hereditary cancer genetic screening and testing in primary care. The total costs for each arm are presented in outcome 3 above. The incremental cost is the difference in total costs when comparing the DPE arm to the POC arm (DPE minus POC).
Time Frame: 2 years
Population: Costs and outcomes were compared between the two arms, with POC as the comparator (standard); that is DPE minus POC. Costs were calculated at the per-patient level and scaled to apply to a theoretical healthcare system with 100,000 patients. As this outcome is the difference between the two strategies, only one value is calculated using the data from the two arms combined. The total costs per arm used for this calculation are shown in outcome 3 above.
Measure: Number; unit: cost in $
Groups:
- Direct Patient Engagement Compared to Point of Care: Clinics in the direct patient engagement (DPE) arm contacted patients by postal mail and email to provide a link to the online familial cancer risk screening tool.
  Clinics in the point of care (POC) arm approached patients at the time they came in to the clinic for a routine visit with their primary care provider.
  The two arms are combined for this analysis.
Arm/Group | Direct Patient Engagement Compared to Point of Care
Number analyzed (Participants) | 51,319
cost in $
  Incremental cost from health-system perspective | 56,340
  Incremental cost from limited societal perspective (includes patient costs) | 49,955

5. Secondary Outcome: Rates of Screening and Testing at Healthcare System A
Description: The table displays the percentages (i.e., proportions) of screening and testing that occurred in the study. The number of patients screened and the number tested are listed as well, but as the denominators differ, the results for Outcome 6 will be based on scaling the proportions to a theoretical healthcare system with 100,000 patients. This information will then be used along with the incremental costs for a healthcare system with 100,000 patients (Outcome 4) to determine the incremental cost-effectiveness ratios (ICERs) presented in Outcome 7.
Time Frame: 2 years
Population: Data from only one of the participating healthcare systems were used. There were 3 clinics in the POC arm and 3 clinics in the DPE arm. The percentages (i.e. proportions) in the table are based on study participant counts. These proportions will be scaled to a healthcare system of 100,000 patients when calculating the incremental differences for Outcome 6.
Measure: Count of Participants; unit: Participants
Arm/Group | Point of Care | Direct Patient Engagement
Number analyzed (Participants) | 29,862 | 21,457
Participants
  Patients screened | 4,327 | 1,370
  Patients tested | 233 | 254

6. Secondary Outcome: Incremental Patients Screened; Incremental Patients Tested
Description: This outcome is the comparative (incremental) difference between the two different engagement strategies in screening and testing outcomes. The total patients screened and tested for each arm are presented in outcome 5 above. The proportions for these outcomes were then scaled to a healthcare system of 100,000 patients and the incremental difference was calculated by comparing the DPE arm to the POC arm (DPE minus POC). Scaling the numbers to a healthcare system of 100,000 patients is necessary for this component to be compatible with the costs for a healthcare system of 100,000 patients given in Outcome 4, in order to calculate the ICERs (Outcome 7).
Time Frame: 2 years
Population: NOTE: percentages (i.e., proportions) shown in Outcome 5 were scaled to a healthcare system of 100,000 patients before calculating these incremental differences. Outcomes were then compared between the two arms (DPE minus POC). As this outcome is the difference between the two strategies, only one value is calculated using the data from the two arms combined. Again, differences were calculated after scaling the proportions, rather than simply using the participant counts from Outcome 5.
Measure: Number; unit: participants
Arm/Group | Direct Patient Engagement Compared to Point of Care
Number analyzed (Participants) | 51,319
participants
  Incremental patients screened | -8,105
  Incremental patients tested | 404

7. Secondary Outcome: Incremental Cost-effectiveness Ratio (ICER) Per Patient Screened; Incremental Cost-effectiveness Ratio Per Patient Tested
Description: This outcome is the Incremental Cost-effectiveness Ratio (ICER). The ICER estimates how much the DPE strategy costs, relative to the POC strategy (DPE minus POC), to improve the outcome measure by 1 unit (in this case one additional patient screened or one additional patient tested). The ICER is calculated by using the difference in costs (outcome 4) divided by the difference in outcome (outcome 6). When the numerator is positive and the denominator is negative (as it is for screening), general practice is to state the second strategy (DPE in this case) was "dominated" by the first strategy (the standard, which is POC in this case). A negative ICER can be misinterpreted, making this clarification necessary.
Time Frame: 2 years
Population: Costs and outcomes were compared between the two arms, with POC as the comparator (standard); in other words DPE minus POC. This combination of the two arms was the prespecified analysis. Cost effectiveness was calculated at the per-patient level, then scaled to apply to a theoretical healthcare system with 100,000 patients.
Measure: Number; unit: $ per additional patient
Arm/Group | Direct Patient Engagement Compared to Point of Care
Number analyzed (Participants) | 51,319
$ per additional patient
  ICER per additional patient screened from health-system perspective | -7
  ICER per additional patient screened from limited societal perspective | -6
  ICER per additional patient tested from health-system perspective | 140
  ICER per additional patient tested from limited societal perspective | 124

ADVERSE EVENTS:
Description: Adverse events were not assessed for any arm in this study, as study activities consisted of surveys and interviews. Genetic testing was offered to eligible patients as standard of care.
Arm/Group | Point of Care | Direct Patient Engagement
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic affected the study as a whole, and the POC arm in particular. One of the healthcare systems shut down clinic waiting rooms and converted most appointments to telehealth. As a result, half of the POC clinics pivoted to telephone engagement. In the remaining POC clinics, genetic testing kits were not handed to eligible patients at the time the patient was found to be eligible, due to COVID precautions and time constraints in-clinic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-16): https://cdn.clinicaltrials.gov/large-docs/94/NCT04746794/Prot_SAP_000.pdf